CLINICAL TRIAL: NCT04271241
Title: Evidence of Central and Local Vascular Function Improvements After Chronic Passive Stretching
Brief Title: Vascular Function Improvements After Chronic Passive Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Emilano Cè, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stretching vasomotor response
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Vasodilation; Vasoconstriction; Stretch; Sympathetic; Imbalance
Keywords: Chronic passive stretching; Central and peripheral arterial stiffness; Blood pressure; Vasomotor response; Crossover effect
MeSH Terms: conditions — Aneurysm | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Four groups in parallel (three intervention groups and one control) tested at the beginning, during, after and after six weeks (follow-up) from intervention
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor are in-blind about the participants' allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Ctrl) (No Intervention): Ctrl group di not undergo any training
- PS bilateral limbs (PSBil) (Experimental): PSBil underwent 12 weeks of passive stretching on both the lower limbs
  Interventions: Other: Passive stretching (PS) training
- PS monolateral limb, stretched limb (PSMonoSL) (Experimental): PSMonoSL underwent 12 weeks of passive stretching on just one lower limb (SL). Outcomes form this group were obtained from the stretched
  Interventions: Other: Passive stretching (PS) training
- PS monolateral limb, contralateral limb PSMonoCL (Experimental): PSMonoCL involved the same participants as in PSMonoSL. Outcomes form this group were obtained from the contralateral not stretched limb (CL). Data from this limb helped in identify possible PS-induced crossover effects in the vasomotor response.
  Interventions: Other: Passive stretching (PS) training

INTERVENTIONS:
Other: Passive stretching (PS) training — PSBil and PSMono underwent 12 weeks of PS training, 3 sessions per week (36 sessions in total). In PSBil, each session lasted 40 min and included two maneuvers for both the knee extensor and plantar flexor muscles with the following protocol: 45 s elongation and 15 s recovery in the resting position, all the cycle repeated for five times 7. In PSMono, exercises were performed only on the right limb and each session had a duration of 20 min. Ctrl did not underwent any PS exercise throughout the study. To promote participants' compliance, daily classes were held at different day time (morning and afternoon) at the University Sports Centre gym. Each class was supervised by an expert operator, which monitored the attendance, the correct exercise execution and the intensity exerted during the exercise (80% of the point of discomfort). The participants not attending at least the 80% of classes were excluded from the study, and a new participant was recruited to substitute the drop out.
  Arms: PS bilateral limbs (PSBil); PS monolateral limb, contralateral limb PSMonoCL; PS monolateral limb, stretched limb (PSMonoSL)

SUMMARY:
Acutely, during different bouts of passive stretching (PS), blood flow (Q ̇) and shear rate ( ) in the feeding artery of the stretched muscles increases during the first two elongations and then it reduces during the following bouts. This hyperemic response during the first two elongations is mediated by the local release of vasoactive molecules (e.g. nitric oxide, NO). This phenomenon disappears during the following elongations due to the NO and other vasoactive molecule depletion. The relaxation phase between stretching bouts, instead, is always characterized by hyperemia as results of stretch-induced peripheral resistances decrease. Whether chronic PS administration may influence vascular function is still a matter of investigation. The hypothesis is that repetitive PS-induced Q ̇ and changes may be an enough stimulus to provoke increments in NO bioavailability, thus improving vasomotor response.

DETAILED DESCRIPTION:
Vasomotor response is an important marker of cardiovascular health and has been related to cardiovascular co-morbidity. An alteration of vasomotor response, indeed, often precedes an increase in arterial stiffness. By improving and/or maintaining this vascular function, therefore, plays a pivotal role in the prevention of cardiovascular disease. The overall control of the vasomotor response and, in turn, of blood flow distribution in the human body is regulated by two main mechanisms: a systemic control given by the sympathetic nervous system that acts on the arterial smooth muscle fibers causing vasoconstriction, and a local action of vasoactive molecules released by the endothelial cells, such as nitric oxide (NO), leading to vasodilation.

Recent studies report that acute passive stretching (PS), a well-established practice in rehabilitation and sport environments to increase range of motion, may influence the vasomotor response. Specifically, PS provokes two conflicting events: (i) a vasoconstriction with blood flow reduction in the feeding artery of the stretched muscle, triggered by the systemic increase in sympathetic neural tone due to the PS-induced stress on the muscle mechano- and metaboreceptors, and (ii) a vasodilation and subsequent increase in blood flow in the feeding artery due to the prevalence of local vasoactive factors release as a result of the stretch-induced stress applied to the vessel wall, which overwhelms the systemic sympathetic activation. Interestingly, throughout several stretch-shortening cycles, the first acute hyperemic response to stretch described above seems to progressively attenuate until its disappearance during the subsequent stretching cycles, possibly due to NO and other vasoactive molecules depletion.

The shortening phase in between two stretch bouts, instead, is always characterized by hyperemia due to a reduction in the peripheral vascular resistance after the stretch-induced vessels deformation. Possible explanation of these phenomena involves the shear rate, which is the frictional or drag force acting on the inner lumen of the vessels that can trigger a chain of reactions, possibly leading to higher endothelial NO-synthase activity. Continuous and repetitive increases in shear rate induced by PS have been observed to act as vascular training to modulate endothelium remodeling and to improve vasomotor response.

Interestingly, during an acute PS administration, a reduction in blood flow during stretching was described in the contralateral, no-stretched limb. Such a reduction was promptly recovered during the shortening phase. The authors suggested that this occurrence was induced by a systemic sympathetic-mediated vasoconstriction, which was activated by the stretch-induced mechanoreflex.

However, whether chronic PS administration may also affect the vasomotor response in the feeding artery of the contralateral muscle, which was not directly involved in the stretching maneuver, is still an open question.

Together with the changes in local control mechanisms, also possible PS-induced changes in the systemic autonomic control of blood flow has been reported (i.e., reduction in blood pressure and aortic wave reflection magnitude, although its effectiveness remains a matter of debate With this in mind, this study aimed to investigate the effect of PS on the vasomotor response and the stiffness of the arteries directly involved (i.e., femoral and popliteal arteries) and not directly involved (i.e., contralateral femoral and popliteal arteries and brachial artery) with the maneuver applied on the plantar flexors, knee extensor and hip flexor muscles. To this purpose, vasomotor response and arterial stiffness were assessed by Doppler ultrasounds and applanation tonometry, respectively, before and after 12 weeks of PS administration. Hypothesis has been made that repetitive PS bouts, with consequent changes in blood flow and shear rate, may be an effective stimulus to (i) enhance local vasoactive molecules bioavailability in the arteries involved with PS; and (ii) induce a systemic re-modulation of the sympathetic autonomic activity, thus improving arterial compliance and vasomotor response even in those districts not directly involved with PS.

ELIGIBILITY:
Inclusion criteria:

• None

Exclusion criteria:

* presence of neurological, vascular and musculoskeletal impairments at the lower and upper limbs level;
* being on pharmacological therapy related to either neural and/or vascular response, including hormonal contraceptives and oral supplements;
* being a current or former smoker;
* having an irregular menstrual cycle (26 to 35 days) up to three months before the beginning of the study,
* presenting contraindication for joint mobilization;
* being regularly involved in PS program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in augmentation Index | Change from baseline in Augmentation Index at 12 weeks
  The radial artery pressure wave and amplitude were recorded non-invasively by means of applanation tonometry of the radial artery. Twenty sequential waveforms covering a complete respiratory cycle were acquired from the system and used by the software to generate an average peripheral and corresponding central waveform. The systolic part of the wave form was characterized by two pressure peaks of the central waveform. The first peak results from the left cardiac ventricle ejection while the second one results from the wave reflections from the periphery. The difference between these two peaks represents the degree of the central arterial pressure augmentation due to wave reflection (i.e., the augmentation index, mmHg)
Change from baseline in femoral artery delta blood flow | Change from baseline in Delta Blood Flow at 12 weeks
  Femoral artery blood flow was calculated by Doppler ultrasound at baseline and at peak after single passive knee flexion and extension by using the femoral artery diameter and mean blood velocity. The difference between baseline and at peak blood flow identifies the Delta Blood Flow (ml/min).
Change from baseline in brachial artery flow mediated dilation | Change from baseline in brachial artery flow mediated dilation at 12 weeks
  Flow mediated dilation was performed at brachial artery level. An arterial pressure cuff was placed around the forearm immediately distal to the olecranon process to provide an ischemic stimulus when inflated. Following baseline assessment, the blood pressure cuff was inflated to 250 mmHg. Artery diameter was and blood flow were resumed at baseline, 30 s prior to cuff deflation and continued for 2 min post-deflation by a linear array transducer attached to a high-resolution ultrasound machine. When an optimal image was obtained, the probe was held stable and longitudinal in B-mode, acquiring images of the lumen-arterial wall interface. Continuous Doppler velocity assessments were also obtained and collected using the lowest possible insonation angle (<60°). Data were exported and analyzed using commercially available software. Flow mediated dilation was quantified as the maximal change in artery diameter after cuff release, expressed as a percentage increase above baseline (%).

SECONDARY OUTCOMES:
Change from baseline in knee range of motion | Change from baseline in in Knee Range of Motion at 12 weeks
  To monitor the changes in knee range of motion, a bi-axial electrogoniometer was utilized. For the knee joint, the electrogoniometer was placed with one axis on the external condyle of the knee and the other on the external face of the fibula. The knee range of motion was expressed in degrees (deg)
Change in knee extensor muscles maximum isometric voluntary contraction | Before, after 6 weeks, at the end (12th week), and after 6 weeks (Follow-up) of PS training
  The maximum isometric voluntary contraction of the knee extensor muscles was measured with the participant laying supine on an ergometer with the knee flexed at 90° and firmly secured at the ankle level by a Velcro® strap to a load cell for the force signal detection. Hip and shoulders were also firmly secured to the ergometer. After a warm-up (10 x 2-s contractions at 50% maximum isometric voluntary contraction), three maximum isometric voluntary contraction attempts were performed, interspersed by at least 3 min of recovery. The participants were instructed to push as fast and hard as possible for 3 s. The maximum isometric voluntary contraction (N) was identified as the highest force produced during contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Cè, PhD, Principal Investigator — University of Milan
Locations (1):
- Department of Biomedical Science for Health, Milan, Italy